CLINICAL TRIAL: NCT05809297
Title: Diode Laser and Photodynamic Therapy Versus Ciclopirox Hydroxypropyl Chitosan. Randomised Controlled Clinical Trial.
Brief Title: Diode Laser and Photodynamic Therapy Vs. Ciclopirox.
Acronym: Laser
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, FRANCISCO JAVIER ALVARO AFONSO, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nº EudraCT 2022-003913-12
Record Dates: First submitted 2023-03-15; First posted 2023-04-12 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Onychomycosis
Keywords: onychomycosis; laser; ciclopirox
MeSH Terms: conditions — Onychomycosis | interventions — Lasers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Diode laser combined with photodynamic-red laser therapy by RapidoPodia Laser Diodo® (MEDENCY) (Experimental): According to the manufacturer's recommendations, the treatment will be carried out in consultation in 8 sessions by a specialised podiatrist.
  Interventions: Device: Diode laser combined with photodynamic-red laser therapy by RapidoPodia Laser Diodo®
- Ciclopirox Hydroxypropyl Chitosan (HPCH) Nail Lacquer (Active Comparator): The application of Ciclopirox Hydroxypropyl Chitosan (HPCH) Nail Lacquer will be performed at home by the patient once a day.
  Interventions: Drug: Ciclopirox Hydroxypropyl Chitosan (HPCH) Nail Lacquer

INTERVENTIONS:
Device: Diode laser combined with photodynamic-red laser therapy by RapidoPodia Laser Diodo® — According to the manufacturer's recommendations, the treatment will be carried out in consultation in 8 sessions by a specialised podiatrist.
  Other Names: Laser
  Arms: Diode laser combined with photodynamic-red laser therapy by RapidoPodia Laser Diodo® (MEDENCY)
Drug: Ciclopirox Hydroxypropyl Chitosan (HPCH) Nail Lacquer — The application of Ciclopirox Hydroxypropyl Chitosan (HPCH) Nail Lacquer will be performed at home by the patient once a day.
  Other Names: Control
  Arms: Ciclopirox Hydroxypropyl Chitosan (HPCH) Nail Lacquer

SUMMARY:
The main objective of this study is to compare the efficacy of treatment of onychomycosis by: diode laser combined with photodynamic therapy, and topical treatment with Ciclopirox Hydroxypropyl Chitosan (HPCH) Nail Lacquer.

The study is a low-intervention, randomised controlled clinical trial. Patient recruitment will be done by including in the sample those patients who have diagnostic confirmation of onychomycosis in the Chiropodology and Surgery Service of the University Podiatry Clinic of the Complutense University of Madrid. Participants in the trial will be assigned with equal probability to each treatment arm, according to their consecutive inclusion in the study. Subsequently, treatment assignment will be determined by a random code. The treatment used will be evident to both the participant and the podiatrist responsible for the intervention.

Visits will be made every 7 days at the start of treatment and for 9 weeks in group 1 (treatment with laser and photodynamic therapy), and monthly visits in group 2 (treatment with ciclopirox nail polish) during the 12 months of follow-up. Regardless of the follow-up week at which healing occurs, all patients will be reviewed at 3, 6, 9 and 12 months after the first visit.

DETAILED DESCRIPTION:
Visits will be made every 7 days at the start of treatment and for 9 weeks in group 1 (treatment with laser and photodynamic therapy), and monthly visits in group 2 (treatment with ciclopirox nail polish) during the 12 months of follow-up. Regardless of the follow-up week at which healing occurs, all patients will be reviewed at 3, 6, 9 and 12 months after the first visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with toenail onychomycosis with positive microbiological culture/PCR.
* Patients over 18 years of age.

Exclusion Criteria:

* Patients who have received topical or systemic antifungal treatment in the previous month.
* Pregnancy or lactation.
* Patients with peripheral vascular disease.
* Patients with an immune system disorder or undergoing treatment with immunosuppressants.
* Patients with peripheral or central neuropathy.
* Patients with a coagulation disorder.
* Patients with Raynaud's disease or with any alteration in the perception of cold or heat.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of treatment of onychomycosis with diode laser combined with photodynamic therapy versus Ciclopirox Hydroxypropyl Chitosan (HPCH) Nail Lacquer. | 12 months
  Clinical cure (yes/no).
Efficacy of treatment of onychomycosis with diode laser combined with photodynamic therapy versus Ciclopirox Hydroxypropyl Chitosan (HPCH) Nail Lacquer. | 12 months
  Mycological cure (yes/no)
Efficacy of treatment of onychomycosis with diode laser combined with photodynamic therapy versus Ciclopirox Hydroxypropyl Chitosan (HPCH) Nail Lacquer. | 12 months
  Complete cure (yes/no)

SECONDARY OUTCOMES:
To determine whether 8 sessions of diode laser treatment combined with photodynamic therapy, at different wavelengths, over a period of nine weeks, is sufficient to achieve clinical cure of onychomycosis. | 12 months
  Clinical cure (yes/no)
To determine whether 8 sessions of diode laser treatment combined with photodynamic therapy, at different wavelengths, over a period of nine weeks, is sufficient to achieve, mycological cure of onychomycosis. | 12 months
  Mycological cure (yes/no).
To determine whether 8 sessions of diode laser treatment combined with photodynamic therapy, at different wavelengths, over a period of nine weeks, is sufficient to achieve complete cure of onychomycosis. | 12 months
  Complete cure (yes/no).
To analyse the influence of the type of onychomycosis on the response to treatment. | 12 months
  Onychomycosis clasification (ODL, total dystrophic, superficial)
To analyse the influence of the causal fungal agent on the response to treatment. | 12 months
  Causal fungal agent (dermatophyte, mould or yeast)
To analyse the influence of the degree of severity of onychomycosis on the response to treatment. | 12 months
  Onychomycosis severity index (OSI)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Álvaro Afonso, Principal Investigator — Universidad Complutense de Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Oreja S, Alvaro-Afonso FJ, Navarro-Perez D, Leon-Herce D, Tardaguila-Garcia A, Lazaro-Martinez JL. Diode Laser and Red-Laser Photodynamic Therapy Versus Ciclopirox 8% HPCH Nail Lacquer for the Treatment of Onychomycosis: A Randomised Controlled Trial. Mycoses. 2025 Oct;68(10):e70121. doi: 10.1111/myc.70121. PMID 41024682